CLINICAL TRIAL: NCT01878110
Title: Treatment Development Study of the COMB Model of Trichotillomania
Brief Title: Efficacy of COMB (Comprehensive Behavioral) Model of Treatment of Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: Trichotillomania Learning Center (Other)
Responsible Party: Principal Investigator, David A. F. Haaga, Professor of Psychology, American University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLC COMB Pilot Study; TLC (Other Grant/Funding Number: Trichotillomania Learning Center)
Record Dates: First submitted 2013-06-10; First posted 2013-06-14 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Trichotillomania; Hair-Pulling Disorder
Keywords: Trichotillomania; Hair pulling; Behavior therapy
MeSH Terms: conditions — Trichotillomania

ARMS (1):
- COMB (Experimental)
  Interventions: Behavioral: COMB

INTERVENTIONS:
Behavioral: COMB

SUMMARY:
This pilot study is being conducted in order to help make the case for later, more systematic research on the effectiveness of the Comprehensive Behavioral (COMB) model of treating trichotillomania (compulsive hair pulling). The goals are to standardize COMB treatment techniques in the form of a clear written manual for therapists; determine whether therapists can use these guidelines in a consistent manner in making treatment decisions; develop and test the reliability of measures of how well therapists are conducting the treatment; and collect preliminary data on the acceptability of the treatment to patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary Diagnostic and Statistical Manual, Fifth Edition (DSM-5) diagnosis of Trichotillomania (TTM)

Exclusion Criteria:

* Current suicidality or severe depression
* Current psychosis
* Current alcohol or substance abuse
* Concurrent psychotherapy for TTM
* Psychotropic meds (for any disorder) that have not been stable for >4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Massachusetts General Hospital Hairpulling Scale (MGH-HS) | 12 weeks
  Improvement in hair pulling symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States